CLINICAL TRIAL: NCT00472589
Title: A Biological Sample Collection Protocol of Women With and Without Breast Cancer: Hoosier Oncology Group Study BRE06-120 for the Analytical Proteomics Team
Brief Title: A Biological Sample Collection Protocol of Women With and Without Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: Purdue University (Other); Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: BRE06-120; BRE06-120 (Registry Identifier: ClinicalTrials.Gov)
Record Dates: First submitted 2007-05-09; First posted 2007-05-11 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, serum, whole blood and tissue samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Healthy women
- 2: Women with breast cancer

SUMMARY:
The purpose of this trial is to collect plasma, serum, whole blood and tissue samples from women with breast cancer and plasma, serum, whole blood from healthy women, which will be made available to researchers for biomarker analysis.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

The treatment plan for each breast cancer subject will be determined at the discretion of the treating physician and subject. This protocol does not prescribe any particular standard of care treatment.

There will be no treatment for the healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

FOR WOMEN WITH BREAST CANCER

* Histologically or cytologically confirmed invasive malignancy or ductal carcinoma in situ of the breast.
* Preparing to begin a new regimen for breast cancer (adjuvant, locally recurrent, any line metastatic).
* Female.
* Age > 18 years at the time of consent.
* Written informed consent and HIPAA authorization for release of personal health information.

FOR HEALTHY VOLUNTEERS

* No known history of invasive malignancy or ductal carcinoma in situ. Volunteers must not have prior history of malignancy in the past 5 years with the exception of basal cell and squamous cell carcinoma of the skin. Other cancers with low potential for metastasis, such as in situ cancers (e.g., Grade 1, TA TCC (low grade superficial bladder cancer), colonic polyp with focus of adenocarcinoma) can also be enrolled as healthy volunteers.
* Female
* Age > 18 years at the time of consent.
* Written informed consent and HIPAA authorization for release of personal health information.

Exclusion Criteria:

* Females must not be pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy women and women with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2007-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Schneider, M.D., Study Chair — Hoosier Oncology Group, LLC; Fred Regnier, Principal Investigator — Purdue University
Locations (11):
- United States (11):
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Cancer Care Center of Southern Indiana, Bloomington, Indiana
  - Oncology Hematology Associates of SW Indiana, Evansville, Indiana
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Quality Cancer Center (MCGOP), Indianapolis, Indiana
  - Arnett Cancer Care, Lafayette, Indiana
  - Horizon Oncology Center, Lafayette, Indiana
  - Medical Consultants, P.C., Muncie, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Oncology Partners Network, Cincinnati, Ohio

REFERENCES:
- See also: Hoosier Oncology Group Homepage — http://www.hoosieroncologygroup.org